CLINICAL TRIAL: NCT06825520
Title: Investigating Changes in Premonitory Urges During Habit Reversal Training
Brief Title: Investigating Changes in Premonitory Urges During Habit Reversal Training for Tics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Emily Braley, University of Utah, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00183697
Record Dates: First submitted 2025-02-05; First posted 2025-02-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Tics; Tourette Disorder; Tourette Syndrome in Children; Tourette Syndrome in Adolescence
Keywords: habit reversal training; tics; tourette; tourette's disorder; Tourette syndrome; treatment for tics
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRT (Experimental): Participants will receive 3 therapist-guided sessions of habit reversal training (1 hour each) for 3 separate identified tics. Participant will also participate in 5 practice sessions per week (approximately 30 minutes sessions each; over the course of 3 weeks) in which participants will practice the skills learned in session with a study team member)
  Interventions: Behavioral: Habit Reversal Training

INTERVENTIONS:
Behavioral: Habit Reversal Training — Participants learn to identify when their tics occur and then learn a competing response to engage in instead of the 3 identified tics and then practice competing responses learned in session during the practice sessions throughout the week.

SUMMARY:
The primary aim of this study is to learn more about premonitory urges (PU) when using Habit Reversal Training (HRT) to treat tics.

The main focus of this study is to investigate if and when PU change during tic treatment sessions and between tic treatment sessions.

Participants will:

* Attend 5 study visits (approximately 1 to 1.5 hours each) for an intake, habit reversal training for 3 separate tics, and a post assessment
* Attend 5 practice sessions (approximately 30 minutes each) over a week for 3 weeks (total 15 practice sessions)
* Study visits and practice sessions will take place in person and online via secure videoconference

DETAILED DESCRIPTION:
Current research has shown that although tics can be effectively reduced with short-term suppression strategies or habit reversal training (HRT), it remains unclear whether improvement in tic symptoms is accompanied by a reduction in premonitory urges (PUs). Premonitory urges are uncomfortable premonitory sensations that signal a tic is about to occur. Most individuals describe these premonitory sensations as an itch, pressure, energy, or other uncomfortable or "not just right" sensation that is usually localized to the area of the body in which the tic occurs. Furthermore, most individuals report that their PUs increase when tics are suppressed and are reduced or eliminated, albeit temporarily, after the tic is executed. Because the execution of tics reduces aversive PUs, it has been hypothesized that they are strengthened, shaped, and maintained, at least in part, by automatic negative reinforcement. Further investigation into the PU-tic association during treatment is needed. A better understanding of how PUs fluctuate during HRT (both within and between sessions) will potentially provide further insight into its underlying mechanism(s). A better understanding of how PUs fluctuate during HRT (both within and between sessions) will potentially provide further insight into its underlying mechanism(s). Specifically, if tics reduce but PU do not reduce when within and between HRT sessions, such findings would cast doubt on the role of habituation and spur the investigation of alternative hypotheses. The primary aim of this study is to contribute to the current literature on the model of tic maintenance and reduction and the PU-tic association by investigating individual PU severity fluctuations within and between sessions when using HRT to treat tics. Specifically, the study will examine whether subjective ratings of PUs decrease within and between sessions following HRT, as would be expected from the habituation hypothesis.

The primary aim of this study is to contribute to the current literature on the model of tic maintenance and reduction and the PU-tic association by investigating individual PU severity fluctuations within and between sessions when using HRT to treat tics.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet criteria for a DSM-5-TR diagnosis of a TD will be recruited to participate in this study. Participants will be eligible for the study if they

1. present with at least three motor and/or vocal tics and are interested in receiving treatment,
2. report experiencing a PU for each of their target tics with a minimum rating of a 4/8 on a subjective rating (i.e., the Urge Thermometer; Silverman & Albano, 1996) for each tic,
3. the targeted tics occur, on average, at least once per minute during a 10-minute direct observation,
4. are between the ages of 8 and 17
5. the patient has no planned changes in medication initiation or dosage during their study participation period.

Exclusion Criteria:

1. the presence of any comorbid conditions that are considered a primary treatment concern and/or could interfere with study participation or treatment (i.e., unmanaged ADHD, OCD, anxiety),
2. have previously engaged in CBIT or HRT for more than 2 sessions,
3. a Yale Global Tic Severity Score of 40+ (or 20+ if they present with a primary motor or vocal tic disorder),
4. suspected (based on clinical presentation) that the tics are better attributed to functional neurological symptom disorder per DSM-5-TR criteria (APA, 2022).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Premonitory Urge (PU) Severity as measured by the urge thermometer | PU severity will be measured during a 10 minute baseline observation; approximately 15 minutes or until 5 CR initiations have occurred, whichever is longer during each of the 3 HRT sessions and 15 practice sessions; during the 15 minute post assessment
  Premonitory urge (PU) severity is an subjective measure of PU ratings while participants are implementing their competing response during study treatment sessions or practice sessions. The Urge Thermometer is an adapted version of the "feelings thermometer" from the Anxiety Disorders Interview Schedule for DSM-IV. It is a 9-point rating scale, ranging from 0 to 8 with higher scores indicating stronger urge experiences, designed to efficiently collect the patients' subjective rating of the severity/intensity of their urge.

SECONDARY OUTCOMES:
Tic Change as measured by tic counts | Tics will be counted during a 10 minute baseline observation; approximately 15 minutes or until 5 CR initiations have occurred, whichever is longer during each of the 3 HRT sessions and 15 practice sessions; during the 15 minute post assessment
  Coding for tics will utilize 10-second partial interval coding in which the presence or absence of each target tic is recorded as present or absent in each 10-s interval. Tic rate will be calculated by dividing the number of intervals in which each target tic is present by the total number of intervals and multiplying this number by 100%. Ten-second partial interval coding has been shown to provide a reliable and valid measure of tics over observation periods of 5 minutes or longer (Himle et al., 2006).

OTHER OUTCOMES:
Participant scores on Treatment Expectancy and Acceptability Questionnaire at baseline | Given at baseline (first study visit)
  At the baseline assessment, participants will be asked to rate how much they believe in the treatment on a 5-point scale, and how much they think their tics will improve on a 5-point scale with additional questions from the Credibility/Expectancy Questionnaire (Devilly & Borkovec, 2000). Scores can range from 3 to 15. Participants will also be asked to rate treatment acceptability at pre-treatment (including questions about the acceptability, ethicality, effectiveness, and potential negative side effects of the treatment). Questions are rated on a 1 to 7 scale, with lower scores representing more negative impressions and reactions to the proposed treatment. Scores can be totaled ranging from 6 to 42.
Patient scores on Satisfaction with Therapy and Therapist Scale- Revised (STTS-R) post treatment | Given at post assessment (final study visit) approximately 5 weeks from study initiation
  The STTS is a commonly used 13-item self-report measure that assesses patients' satisfaction with their therapist and the treatment that they received. Each item is rated on a 5-point Likert-type scale with higher scores indicating greater overall satisfaction with treatment and the therapist. Scores range from 15 to 65.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in any publication(s) may be provided to qualified researchers. All data shared will be coded with no identifying information included. Approval of the request by the study primary investigator and execution of all applicable data sharing agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication.
Access Criteria: Qualified researchers are those considered to have academic interests in tic disorders and related conditions, expertise in the scoring and interpretation of the outcome measures administered, and a reasonable and scientifically-sound justification for obtaining participant data.

REFERENCES:
- [Background] Woods DW, Walther MR, Bauer CC, Kemp JJ, Conelea CA. The development of stimulus control over tics: a potential explanation for contextually-based variability in the symptoms of Tourette syndrome. Behav Res Ther. 2009 Jan;47(1):41-7. doi: 10.1016/j.brat.2008.10.013. Epub 2008 Oct 21. PMID 19026406
- [Background] Woods DW, Piacentini JC, Scahill L, Peterson AL, Wilhelm S, Chang S, Deckersbach T, McGuire J, Specht M, Conelea CA, Rozenman M, Dzuria J, Liu H, Levi-Pearl S, Walkup JT. Behavior therapy for tics in children: acute and long-term effects on psychiatric and psychosocial functioning. J Child Neurol. 2011 Jul;26(7):858-65. doi: 10.1177/0883073810397046. Epub 2011 May 9. PMID 21555779
- [Background] Wilhelm S, Deckersbach T, Coffey BJ, Bohne A, Peterson AL, Baer L. Habit reversal versus supportive psychotherapy for Tourette's disorder: a randomized controlled trial. Am J Psychiatry. 2003 Jun;160(6):1175-7. doi: 10.1176/appi.ajp.160.6.1175. PMID 12777279
- [Background] Wellen BCM, Ramanujam K, Lavelle M, Capriotti MR, Butner J, Euler MJ, Himle MB. A Test of the Behavioral Model of Tic Disorders Using a Dynamical Systems Framework. Behav Ther. 2024 May;55(3):513-527. doi: 10.1016/j.beth.2023.08.010. Epub 2023 Sep 4. PMID 38670665
- [Background] Tolin DF, Sain KS, Davis E, Gilliam C, Hannan SE, Springer KS, Stubbing J, George JR, Jean A, Goldblum R, Katz BW, Everhardt K, Darrow S, Ohr EE, Young ME, Serchuk MD. The DIAMOND-KID: Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders in Children and Adolescents. Assessment. 2023 Dec;30(8):2351-2363. doi: 10.1177/10731911221143994. Epub 2023 Jan 11. PMID 36632642
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] McGuire JF, McBride N, Piacentini J, Johnco C, Lewin AB, Murphy TK, Storch EA. The premonitory urge revisited: An individualized premonitory urge for tics scale. J Psychiatr Res. 2016 Dec;83:176-183. doi: 10.1016/j.jpsychires.2016.09.007. Epub 2016 Sep 9. PMID 27643476
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Houghton DC, Capriotti MR, Scahill LD, Wilhelm S, Peterson AL, Walkup JT, Piacentini J, Woods DW. Investigating Habituation to Premonitory Urges in Behavior Therapy for Tic Disorders. Behav Ther. 2017 Nov;48(6):834-846. doi: 10.1016/j.beth.2017.08.004. Epub 2017 Aug 10. PMID 29029679
- [Background] Himle MB, Woods DW, Conelea CA, Bauer CC, Rice KA. Investigating the effects of tic suppression on premonitory urge ratings in children and adolescents with Tourette's syndrome. Behav Res Ther. 2007 Dec;45(12):2964-76. doi: 10.1016/j.brat.2007.08.007. Epub 2007 Aug 10. PMID 17854764
- [Background] Himle MB, Chang S, Woods DW, Pearlman A, Buzzella B, Bunaciu L, Piacentini JC. Establishing the feasibility of direct observation in the assessment of tics in children with chronic tic disorders. J Appl Behav Anal. 2006 Winter;39(4):429-40. doi: 10.1901/jaba.2006.63-06. PMID 17236340
- [Background] Himle MB, Capriotti MR, Hayes LP, Ramanujam K, Scahill L, Sukhodolsky DG, Wilhelm S, Deckersbach T, Peterson AL, Specht MW, Walkup JT, Chang S, Piacentini J. Variables Associated With Tic Exacerbation in Children With Chronic Tic Disorders. Behav Modif. 2014 Mar;38(2):163-83. doi: 10.1177/0145445514531016. Epub 2014 Apr 28. PMID 24778433
- [Background] Kane MJ. Premonitory urges as "attentional tics" in Tourette's syndrome. J Am Acad Child Adolesc Psychiatry. 1994 Jul-Aug;33(6):805-8. doi: 10.1097/00004583-199407000-00005. PMID 8083137
- [Background] Espil FM, Woods DW, Specht MW, Bennett SM, Walkup JT, Ricketts EJ, McGuire JF, Stiede JT, Schild JS, Chang SW, Peterson AL, Scahill L, Wilhelm S, Piacentini JC. Long-term Outcomes of Behavior Therapy for Youth With Tourette Disorder. J Am Acad Child Adolesc Psychiatry. 2022 Jun;61(6):764-771. doi: 10.1016/j.jaac.2021.08.022. Epub 2021 Sep 8. PMID 34508805
- [Background] Crossley E, Seri S, Stern JS, Robertson MM, Cavanna AE. Premonitory urges for tics in adult patients with Tourette syndrome. Brain Dev. 2014 Jan;36(1):45-50. doi: 10.1016/j.braindev.2012.12.010. Epub 2013 Jan 29. PMID 23369830
- [Background] Capriotti MR, Piacentini JC, Himle MB, Ricketts EJ, Espil FM, Lee HJ, Turkel JE, Woods DW. Assessing Environmental Consequences of Ticcing in Youth with Chronic Tic Disorders: The Tic Accommodation and Reactions Scale. Child Health Care. 2015;44(3):205-220. doi: 10.1080/02739615.2014.948164. Epub 2014 Dec 9. PMID 27076696
- [Background] Capriotti MR, Brandt BC, Turkel JE, Lee HJ, Woods DW. Negative Reinforcement and Premonitory Urges in Youth With Tourette Syndrome: An Experimental Evaluation. Behav Modif. 2014 Mar;38(2):276-96. doi: 10.1177/0145445514531015. Epub 2014 Apr 21. PMID 24752420
- [Background] Capriotti MR, Brandt BC, Ricketts EJ, Espil FM, Woods DW. Comparing the effects of differential reinforcement of other behavior and response-cost contingencies on tics in youth with Tourette syndrome. J Appl Behav Anal. 2012 Summer;45(2):251-63. doi: 10.1901/jaba.2012.45-251. PMID 22844135
- [Background] American Psychiatric Association. (2022). Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revision (DSM-5-TR). American Psychiatric Association Publishing. https://doi.org/10.1176/appi.books.9780890425787